CLINICAL TRIAL: NCT05551624
Title: Evaluation of the Effect in Platelet Count of Atorvastatin and N-acetyl Cysteine in Patients With Primary Immune Thrombocytopenia Resistant to Steroid Treatment or in Relapse: An Exploratory Clinical Trial
Brief Title: Evaluation of the Effect in Platelet Count of Atorvastatin and N-acetyl Cysteine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Enrique Cervantes-Perez, Attending Internal Medicine Physician and Professor to the Department of Internal Medicine, Hospital Civil de Guadalajara "Fray Antonio Alcalde"., Hospital Civil de Guadalajara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 178/19
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: Immune thrombocytopenia; Atorvastatin; N-acetylcysteine; Steroids
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Atorvastatin; Tablets; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Prospective, single group, exploratory (proof of concept) clinical trial to evaluate the effect in serum platelet count of Atorvastatin plus N-acetylcysteine in patients with primary immune thrombocytopenia resistent to steroid therapy or in relapse
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atorvastatin + N-acetylcysteine (Experimental): Patients included in the study received an oral treatment of Atorvastatin 40 mg daily and N-acetylcysteine 400 mg every 8 hours, for at least 1 month (up to 12 months)
  Interventions: Drug: Atorvastatin 40 Mg Oral Tablet + N-acetylcysteine 400 mg Oral tablet

INTERVENTIONS:
Drug: Atorvastatin 40 Mg Oral Tablet + N-acetylcysteine 400 mg Oral tablet — Oral tablets administered daily, atorvastatin once a day and N-acetylcysteine every 8 hours

SUMMARY:
The purpose of this study is to assess the ability of Atorvastatin and N-acetyl cysteine to elevate the blood (serum) platelet count in patients with Immune Thrombocytopenia as a mean of a new treatment.

DETAILED DESCRIPTION:
Evaluate the efficacy in the elevation of platelet count of the combination of atorvastatin and N-acetyl cysteine in patients with immune thrombocytopenia resistant to steroid therapy or with relapse after treatment, a prospective, proof of concept clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients that give their informed consent before the procedures of study
* Thrombocytopenia before intervention (<100 x10^9 /L)
* Patients of either biological sex older than 15 years old
* Patients with previous diagnosis of primary immune thrombocytopenia that not reach complete remission after treatment (steroid based) or that have a relapse
* If the patient is taking steroid based treatment, the dose need to be stable before intervention.

Exclusion Criteria:

* Patients with secondary immune thrombocytopenia
* Pregnant patients
* Patients with hypersensitivity to study treatments
* Patients that are taking anticoagulant medication or any drug that have an effect on platelet count
* Hepatic alteration consisting in serum levels of Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 3 times above superior laboratory reference limit.
* Elevation of serum levels of Creatinine or bilirubins above 1.5 mg/dl
* Any cancer diagnosis
* Coronary heart disease, congestive heart failure, uncontrolled hypertension or arrhythmias.
* Previous autoimmune disease diagnosis including: systemic lupus erythematosus, rheumatoid arthritis or systemic sclerosis.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-04 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2020-01-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline (before intervention) in the Mean Serum Platelet Count at 1, 3, 6 and 12 Months | Baseline and 1, 3, 6, and 12 months after intervention
  Blood samples of all participants will be taken previous to the intervention of study and in the 1, 3, 6, adn 12 month, this with the objective of evaluate changes in platelet count after intervention expecting to elevate the platelet count.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Cervantes-Perez, MD, MSc, Principal Investigator — Hospital Civil de Guadalajara
Locations (1):
- Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco, Mexico